CLINICAL TRIAL: NCT02873247
Title: Prospective Analysis of the Eradication Percentage of Helicobacter Pylori, to Evaluate the Effect of Standardized Eradication Schemes and Active Communication With the General Practitioner and Patient.
Brief Title: Standardize Communication With General Practitioner & Patient for Improved Eradication of Helicobacter Pylori
Acronym: Helipro
Status: Completed | Type: Observational
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Didier Baert, M.D., Algemeen Ziekenhuis Maria Middelares
Other Study IDs: Helipro
Record Dates: First submitted 2015-09-21; First posted 2016-08-19 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients who test Helicobacter pylori positive, are treated with antibiotics. However, due to a number of factors (such as unknown treatment compliance, no standardized follow-up, ...), a relative low eradication-percentage was reported.

Therefore, the investigators want to measure the anticipated improvement in eradication-percentage due to the standardized treatment schedules (1st line, 2nd line and further) and the optimized communication with the general practitioner and patients.

DETAILED DESCRIPTION:
Patients who test Helicobacter pylori positive, are treated with antibiotics. However, due to a number of factors (such as unknown treatment compliance, no standardized follow-up, ...), a relative low eradication percentage was reported. Therefore, the investigators want to measure the anticipated improvement in eradication percentage due to the standardized treatment schemes (1st line, 2nd line and further) and the optimized communication with the general practitioner and patients.

If a patient is eligible (Helicobacter pylori positive) :

1. The standardized eradication scheme in 1st line is:

   sequential therapy being the first 5 days (PPI 2x40mg/d + amoxicilline 2x1g/d), followed by 5 days (PPI 2x40mg/d + clarithromycin 2x500mg/d + flagyl 2x500mg/d)
2. A standardized letter is sent to the general practitioner, mentioning the eradication scheme, and the need to test for eradication success after 8 weeks. A copy of this letter is being sent to the patient. An information folder about Helicobacter pylori infection with instructions on what is expected from the patient, is sent to the patient.
3. After 8 weeks, a control helicobacter pylori breath test (An ureum breath test is a type of test performed on air generated from the act of exhalation ; this test is specific to detect Helicobacter pylori) is performed, and a questionnaire is filled in by the patient.
4. If the ureum breath test is positive, a 2nd line treatment is started = tryplera schedule for 10 days (4x3 co/dag + PPI 2x40mg/d) (1 co tryplera contains 140mg bismuthsubcitrate, 125mg metronidazole, 125mg tetracycline hydrochloride)
5. A standardized letter is sent to the general practitioner, mentioning the 2nd line eradication scheme, and the need to test for eradication success after 8 weeks. A copy of this letter is being sent to the patient.
6. After 8 weeks, a control helicobacter pylori breath test is performed, and a questionnaire is filled in by the patient.
7. If the breath test is positive, a 3rd line treatment is started, based on the results of an antibiogram.
8. A standardized letter is sent to the general practitioner, mentioning the 3rd line eradication schedule, and the need to test for eradication success after 8 weeks. A copy of this letter is being sent to the patient.
9. After 8 weeks, a control helicobacter pylori breath test is performed, and a questionnaire is filled in by the patient.

Overall time-frame : a maximum of 100 helicobacter-positive patients will be recruited over a period of 1 year. Included patients are followed up for 30 weeks maximally.

ELIGIBILITY:
Inclusion Criteria:

* positive test result for Helicobacter pylori (either on a Helicobacter pylori ureum breath test, a biopsy or a faeces test)
* 18+

Exclusion Criteria:

* former failure on Helicobacter pylori eradication with antibiotics
* known allergy for amoxicillin, clarithromycin, flagyl or tryplera

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a positive test result for Helicobacter pylori (either on a Helicobacter pylori ureum breath test, a biopsy or a faeces test)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The presence of Helicobacter pylori is measured using a 13C-ureum breath test (performed minimally 8 wks after the eradication scheme with antibiotics) | Each treatment cycle is about 10 weeks per patient. (10 days antibiotics treatment + 8wks waiting time before Helicobacter pylori breath test). Outcome measurement will be tested at week10, 20 or maximally week30 (depending on number of eradications)
  From all included Helicobacter pylori infected patients, a breath test gives a pos/neg result for the presence of Helicobacter pylori. If not successful after a first antibiotics therapy of 10 days, a second-line antibiotics therapy will be initiated, followed by a breath test after minimally 8 weeks. If not successful after a second treatment, a third-line will be started + breath test to test the eradication. Overall, we aim at an eradication percentage of more than 48%.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Baert, MD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium